CLINICAL TRIAL: NCT00962091
Title: An Open-label, Phase 1 Study of the Relative Bioavailability, Food Effect, Safety and Tolerability of MLN8237 in Patients With Advanced Solid Tumors
Brief Title: Study of MLN8237 in Participants With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: C14010; U1111-1187-6657 (Registry Identifier: WHO)
Record Dates: First submitted 2009-08-18; First posted 2009-08-19 (Estimated); Results first posted 2019-03-12 (Actual); Last update posted 2019-03-12 (Actual); Status verified 2019-03

CONDITIONS: Advanced Solid Tumors
Keywords: Drug therapy
MeSH Terms: interventions — MLN 8237

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (7):
- Dose Escalation (Experimental): A single dose of alisertib 15 mg, oral solution (OS) was administered on Day 1, followed by alisertib 40 mg, powder-in-capsule (PIC), orally, twice a day (BID) on Days 3 through 9, followed by a 14-day rest period in Cycle 1 in a 23-day cycle. A single dose of alisertib 50 mg PIC, orally, was administered on Cycle 2 Day 1 followed by alisertib 40 mg on Days 3 through 9, followed by a 14-day rest period in Cycle 2 in a 23-day cycle. Subsequent cycles, alisertib 40 or 50 mg (individual dosage based on tolerability in Cycles 1 and 2), PIC, orally, BID on Days 1 through 7, followed by a 14-day rest period in 21-day cycles until disease progression, occurrence of an unacceptable alisertib-related toxicity, or the start of another anticancer therapy.
  Interventions: Drug: Alisertib
- Part A: Relative Bioavailability OS/PIC (Sequence A) (Experimental): A single dose of alisertib 25 mg, OS, administered on Day 1, followed by alisertib 40 mg PIC, orally, BID on Days 3 through 9, followed by a 14-day rest period in Cycle 1, in a 23-day cycle. A single dose of alisertib 50 mg PIC, orally, administered on Cycle 2 Day 1, followed by alisertib 40 mg, PIC, orally, BID on Days 3 through 9, followed by a 14-day rest period in a 23-day cycle. Subsequent cycles, alisertib 40-50 mg (individual dosage based on tolerability in Cycles 1 and 2), PIC, orally, BID on Days 1 through 7, followed by a 14-day rest period in 21-day cycles until disease progression, occurrence of an unacceptable alisertib-related toxicity, or the start of another anticancer therapy.
  Interventions: Drug: Alisertib
- Part A: Relative Bioavailability PIC/OS (Sequence B) (Experimental): A single dose of alisertib 50 mg, PIC, orally administered on Day 1, followed by alisertib 40 mg, PIC, orally, BID on Days 3 through 9, followed by a 14-day rest period in Cycle 1, in a 23-day cycle. Cycle 2 Day 1 alisertib 25 mg, OS, once on Day 1, followed by alisertib 40 mg, PIC, orally, BID on Days 3 through 9, followed by a 14-day rest period in a 23-day cycle. Subsequent cycles followed by alisertib 40-50 mg (individual dosage based on tolerability in Cycles 1 and 2), PIC, orally, BID on Days 1 through 7, followed by a 14-day rest period in Cycle 3, in 21-day cycles until disease progression, occurrence of an unacceptable alisertib-related toxicity, or the start of another anticancer therapy.
  Interventions: Drug: Alisertib
- Part B: OS Food Effect Fed/Fasted (Sequence A) (Experimental): Alisertib 35 mg (35 mg = relative bioavailability estimate in Part A as dose of OS that was calculated to yield the area under the concentration time curve of a 50-mg PIC dose): A single dose of alisertib 35 mg oral solution (OS), in fed state, administered on Day 1, followed by alisertib 30 mg, OS, BID on Days 3-9, followed by a 14-day rest period in Cycle 1, in a 23-day cycle. Cycle 2 Day 1 alisertib 35 mg administered, OS, in fasted state, once on Day 1, followed by alisertib 30 mg, OS, BID on Days 3-9, followed by a 14-day rest period in a 23-day cycle. Cycle 3 onwards, participants received alisertib 40 mg, PIC, orally, BID on Days 1-7, with dose reduction to 30 mg BID or escalation to 50 mg BID permitted, based on individual tolerance, followed by a 14-day rest period, in 21-day cycles until disease progression, occurrence of an unacceptable alisertib-related toxicity, or the start of another anticancer therapy.
  Interventions: Drug: Alisertib
- Part B: OS Food Effect Fasted/Fed (Sequence B) (Experimental): A single dose of alisertib 35 mg, OS, in fasted state, administered on Day 1, followed by alisertib 30 mg, OS, BID on Days 3-9, followed by a 14-day rest period in a 23-day cycle. Cycle 2 Day 1 alisertib 30 mg, OS administered in fed state, once on Day 1, followed by alisertib 30 mg, OS, BID on Days 3-9, followed by a 14-day rest period in a 23-day cycle. Cycle 3 onwards, participants received alisertib 40 mg PIC, orally, BID on Days 1-7, with dose reduction to 30 mg BID or escalation to 50 mg BID permitted based on individual tolerance, followed by a 14-day rest period in 21-day cycles until disease progression, occurrence of an unacceptable alisertib-related toxicity, or the start of another anticancer therapy.
  Interventions: Drug: Alisertib
- Part C: ECT Food Effect Fed/Fasted (Sequence A) (Experimental): Alisertib 50 mg, enteric-coated tablets (ECT), orally, in fed state, once on Day 1, followed by alisertib 40 mg, ECT, orally, BID on Days 3 through 9, followed by a 14-day rest period in Cycle 1 in a 23-day cycle, followed by alisertib 50 mg, ECT, orally, in fasted state, once on Day 1, followed by alisertib 40 or 50 mg, ECT, orally, BID on Days 3 through 9, followed by a 14-day rest period in Cycle 2 in a 23-day cycle. Cycle 3 onwards, participants were administered alisertib 40 mg BID ECT on Days 1-7 with dose reduction to 30 mg BID or escalation to 50 mg BID permitted based on individual tolerance, followed by a 14-day rest period in 21-day cycles until disease progression, occurrence of an unacceptable alisertib-related toxicity, or the start of another anticancer therapy.
  Interventions: Drug: Alisertib
- Part C: ECT Food Effect Fasted/Fed (Sequence B) (Experimental): Alisertib 50 mg, ECT, orally, in fasted state, once on Day 1, followed by alisertib 40 mg, ECT, BID on Days 3 through 9, followed by a 14-day rest period in Cycle 1 in a 23-day cycle, followed by alisertib 50 mg, ECT, orally, in fed state, once on Day 1, followed by alisertib 40 or 50 mg, ECT, orally, BID on Days 3 through 9, followed by a 14-day rest period in Cycle 2, a 23-day cycle. Cycle 3 onwards participants were administered alisertib 40 mg BID ECT on Days 1-7, with dose reduction to 30 mg BID or escalation to 50 mg BID permitted based on individual tolerance, followed by a 14-day rest period, in 21-day cycles until disease progression, occurrence of an unacceptable alisertib-related toxicity, or the start of another anticancer therapy.
  Interventions: Drug: Alisertib

INTERVENTIONS:
Drug: Alisertib — Alisertib OS Alisertib PIC Alisertib PIC
  Other Names: MLN8237

SUMMARY:
The purposes of this study were to estimate the relative (Rel) bioavailability (BA) of an oral solution (OS) formulation of alisertib in reference to a powder-in-capsule (PIC) formulation, to characterize the effect of food on the single-dose pharmacokinetics (PK) of alisertib OS and enteric-coated tablets (ECT), to characterize the multiple-dose safety, tolerability, and steady-state PK of alisertib administered as an OS, and to characterize the multiple-dose safety and tolerability of alisertib administered as an ECT.

DETAILED DESCRIPTION:
The drug being tested in this study is called alisertib (MLN8237). Alisertib is being tested to treat people who have advanced solid tumors. This study will look at the relative bioavailability (BA) (Part A), food effect and multiple-dose PK and safety of the oral solution (OS) (Part B) and food effect and safety of the enteric-coated tablet (ECT) formulation (Part C).

The study enrolled 53 patients (pts). Prior to initiation of Part A, 4 participants were enrolled in a dose escalation cohort. Participants in the study received:

• Alisertib 15 mg to 50 mg orally In the first 2 cycles of all 3 parts of the study, a single dose of alisertib was administered on Day 1 (PIC or OS in Part A [n=19 pts]; OS, in the fed or fasted state, in Part B [n=6 pts]; ECT, in the fed or fasted state, in Part C [n=24 pts]), In Part A, participants then continued on the PIC formulation at 40 mg BID for 7 days (Days 3 - 9). In Part B, participants continued on the OS formulation at a calculated dose administered BID for 7 days (Days 3 - 9). In Part C, the ECT formulation was continued at 40 mg BID for 7 days (Days 3 - 9); however, dose escalation to 50 mg BID was permitted after Cycle 1 based on tolerability and safety findings in the prior cycles. All participants took doses at a gap of 12 hours each day for 7 days followed by a 14-day rest period in a 21-days cycle for the remaining cycles.

This multi-center trial was conducted in the United States. The overall time to participate in this study was 30 months. Participants made multiple visits to the clinic, and final assessments were performed approximately 30 days after last dose of study drug.

ELIGIBILITY:
Inclusion Criteria:

Each participant must meet all of the following inclusion criteria to be enrolled in the study:

* 18 years or older
* Histologically or cytologically confirmed metastatic and/or advanced solid tumor
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
* Female participants who are post menopausal, surgically sterile, or agree to practice 2 effective methods of contraception or abstain from heterosexual intercourse
* Male participants who agree to practice effective barrier contraception or agree to abstain from heterosexual intercourse
* Voluntary written consent
* Suitable venous access for study-required blood sampling
* Measurable disease
* Recovered from effects of prior antineoplastic therapy
* Meet required entry laboratory and organ function levels

Exclusion Criteria:

Participants meeting any of the following exclusion criteria are not to be enrolled in the study:

* Female participants who are pregnant or lactating
* Serious medical or psychiatric illness that could interfere with protocol completion
* Major surgery within 14 days of first dose of alisertib
* Antineoplastic therapy, radiation therapy or any experimental therapy 21 days prior to first dose of alisertib
* Nitrosoureas or mitomycin-C within 6 weeks before the first dose of alisertib.
* Autologous stem cell transplant within 3 months before the first dose of alisertib, or prior allogeneic stem cell transplant at any time.
* Active infection requiring systemic therapy, or other serious infection
* Inability to swallow oral medication
* Gastrointestinal (GI) disease or GI procedure that could interfere with oral absorption or tolerance of alisertib
* Symptomatic brain metastasis
* Uncontrolled cardiovascular condition
* Diagnosis or treatment of another malignancy within 2 years preceding first dose of study drug except nonmelanoma skin cancer or in situ malignancy completely resected
* Known history of human immunodeficiency virus (HIV) infection, hepatitis B, or hepatitis C
* Lactose-intolerant (Parts A and B only)
* Prior history of metabolic acidosis (Parts A and B only)
* Use of enzyme-inducing antiepileptic drugs such as phenytoin, carbamazepine or phenobarbital, or rifampin, rifabutin, rifapentine or St. John's wort within 14 days prior to the first dose of alisertib
* A medical condition requiring use of pancreatic enzymes; or daily, chronic , or regular use of proton pump inhibitors (PPI); or histamine (H2) receptor antagonists. Participants who intermittently use these medications must meet the following:

  * No use of PPI within 7 days of first dose of alisertib
  * No use of H2 antagonist or pancreatic enzymes within 24 hours of first dose of alisertib
* Participants requiring full systemic anticoagulation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2009-09-25 (Actual); Primary Completion 2011-12-28 (Actual); Study Completion 2014-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director Clinical Science, Study Director — Millennium Pharmaceuticals, Inc.
Locations (1):
- Premiere Oncology, A Medical Corporation, Santa Monica, California, United States

REFERENCES:
- [Derived] Falchook GS, Zhou X, Venkatakrishnan K, Kurzrock R, Mahalingam D, Goldman JW, Jung J, Ullmann CD, Milch C, Rosen LS, Sarantopoulos J. Effect of Food on the Pharmacokinetics of the Investigational Aurora A Kinase Inhibitor Alisertib (MLN8237) in Patients with Advanced Solid Tumors. Drugs R D. 2016 Mar;16(1):45-52. doi: 10.1007/s40268-015-0114-8. PMID 26689566
- [Derived] Falchook GS, Venkatakrishnan K, Sarantopoulos J, Kurzrock R, Mita AC, Fu S, Mita MM, Zhou X, Jung JA, Ullmann CD, Milch C, Rosen LS. Relative bioavailability of a prototype oral solution of the Aurora A kinase inhibitor alisertib (MLN8237) in patients with advanced solid tumors. Int J Clin Pharmacol Ther. 2015 Jul;53(7):563-72. doi: 10.5414/CP202359. PMID 26073352

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 3 investigative sites in the United States from 25 September 2009 to 01 July 2014.
Pre-assignment Details: Participants with a diagnosis of advanced solid tumors were enrolled to receive alisertib in 1 of 4 parts: Dose Escalation, Part A (relative bioavailability), Part B (food effect and multiple-dose pharmacokinetics of alisertib oral solution [OS]), and Part C (food effect and safety of alisertib enteric-coated tablets [ECT]).
Groups:
- Dose Escalation Cohort: A single dose of alisertib 15 mg, oral solution (OS) was administered on Day 1, followed by alisertib 40 mg, powder-in-capsule (PIC), orally, twice a day (BID) on Days 3 through 9, followed by a 14-day rest period in Cycle 1 in a 23-day cycle. A single dose of alisertib 50 mg PIC, orally, was administered on Cycle 2 Day 1 followed by alisertib 40 mg on Days 3 through 9, followed by a 14-day rest period in Cycle 2 in a 23-day cycle. Subsequent cycles, alisertib 40 or 50 mg (individual dosage based on tolerability in Cycles 1 and 2), PIC, orally, BID on Days 1 through 7, followed by a 14-day rest period in 21-day cycles until disease progression, occurrence of an unacceptable alisertib-related toxicity, or the start of another anticancer therapy.
Period: Overall Study
Arm/Group | Dose Escalation Cohort | Part A: Relative Bioavailability OS/PIC (Sequence A) | Part A: Relative Bioavailability PIC/OS (Sequence B) | Part B: OS Food Effect Fed/Fasted (Sequence A) | Part B: OS Food Effect Fasted/Fed (Sequence B) | Part C: ECT Food Effect Fed/Fasted (Sequence A) | Part C: ECT Food Effect Fasted/Fed (Sequence B)
Started | 4 | 9 | 10 | 3 | 3 | 12 | 12
Completed | 3 | 7 | 9 | 2 | 3 | 11 | 11
Not Completed | 1 | 2 | 1 | 1 | 0 | 1 | 1
Not completed — Withdrawal by Subject | 1 | 2 | 1 | 1 | 0 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety population is defined as all participants who receive any amount of alisertib. Efficacy analysis included all participants who had a baseline response assessment and at least one on-study response assessment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Dose Escalation Cohort | Part A: Relative Bioavailability OS/PIC (Sequence A) | Part A: Relative Bioavailability PIC/OS (Sequence B) | Part B: OS Food Effect Fed/Fasted (Sequence A) | Part B: OS Food Effect Fasted/Fed (Sequence B) | Part C: ECT Food Effect Fed/Fasted (Sequence A) | Part C: ECT Food Effect Fasted/Fed (Sequence B) | Total
Number analyzed (Participants) | 4 | 9 | 10 | 3 | 3 | 12 | 12 | 53
Age, Continuous [Mean (Full Range); unit: years] | 58.3 [57 to 59] | 54.6 [20 to 71] | 54.0 [36 to 70] | 51.7 [31 to 64] | 57.7 [53 to 61] | 57.4 [39 to 72] | 55.2 [46 to 69] | 55.5 [20 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 5 | 1 | 1 | 7 | 9 | 28
  Male | 1 | 7 | 5 | 2 | 2 | 5 | 3 | 25
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic or Latino | 0 | 0 | 2 | 0 | 1 | 2 | 1 | 6
  Not Hispanic or Latino | 4 | 9 | 8 | 3 | 2 | 10 | 11 | 47
Race/Ethnicity, Customized [Number; unit: participants]
  White | 4 | 8 | 9 | 3 | 2 | 12 | 11 | 49
  Black or African American | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 3
  Asian | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 4 | 9 | 10 | 3 | 3 | 12 | 12 | 53
Height [Mean (Full Range); unit: cm] — Population: Number analyzed is the number of participants with available Baseline Height data.
  cm
    number analyzed (Participants) | 4 | 9 | 10 | 3 | 3 | 11 | 10 | 50
    (all) | 167.7 [163 to 175] | 172.6 [154 to 185] | 172.8 [160 to 188] | 160.3 [157 to 163] | 169.1 [159 to 182] | 169.2 [159 to 179] | 160.5 [152 to 169] | 167.4 [152 to 188]
Weight [Mean (Full Range); unit: kg] | 72.7 [66 to 80] | 85.5 [68 to 118] | 81.4 [65 to 120] | 66.3 [45 to 99] | 77.7 [59 to 99] | 73.0 [45 to 98] | 66.1 [43 to 101] | 74.7 [43 to 120]
Body Surface Area (BSA) [Mean (Full Range); unit: m^2] — BSA = sqrt [height (cm) x weight (kg)/3600] Population: Number analyzed is the number of participants with available Baseline BSA data.
  m^2
    number analyzed (Participants) | 4 | 9 | 10 | 3 | 3 | 11 | 10 | 50
    (all) | 1.84 [1.7 to 2.0] | 2.02 [1.8 to 2.4] | 1.97 [1.7 to 2.5] | 1.69 [1.4 to 2.1] | 1.90 [1.6 to 2.2] | 1.82 [1.4 to 2.2] | 1.68 [1.4 to 2.1] | 1.85 [1.4 to 2.5]

OUTCOME MEASURES:

1. Primary Outcome: Part A: Dose-normalized Cmax (Maximum Observed Concentration) for Estimation of Relative Bioavailability for Alisertib Oral Solution (OS) Versus Powder in Capsule Formulations (PIC)
Description: Dose normalized Cmax was obtained using Cmax divided by alisertib dose in milligrams to provide values adjusted to a 1 mg alisertib dose.
Time Frame: Cycles 1 and 2 Day 1 predose and at multiple time points (up to 48 hours) postdose, and, if clinically feasible, at the time of a serious or unusual adverse event (AE) that was judged by the investigator to be treatment related.
Population: Pharmacokinetic (PK)-evaluable population including all participants with sufficient dosing and PK data to reliably estimate PK parameters, with data available for analysis. Data for Cycle 1 and Cycle 2 were combined for analyses.
Measure: Mean (Standard Deviation); unit: nM/mg
Groups:
- Part A: Alisertib OS: Alisertib 25 mg, OS, once on Day 1 in Cycle 1 or Cycle 2.
- Part A: Alisertib PIC: Alisertib 50 mg, PIC, orally once on Day 1 in Cycle 1 or Cycle 2.
Arm/Group | Part A: Alisertib OS | Part A: Alisertib PIC
Number analyzed (Participants) | 17 | 18
nM/mg | 58.78 (22.583) | 31.40 (11.404)
Statistical Analysis 1: Comparison: Part A: Alisertib OS vs Part A: Alisertib PIC; Test type: Superiority or Other; Geometric mean ratio = 1.90, 90% CI 2-sided [1.52 to 2.37] — The CIs are calculated for the difference in the LS means of the ln-transformed Day 1 Cmax values (difference=OS-PIC). Antilogs of the confidence limits for the difference are taken to construct the CIs for the ratio of the geometric means

2. Primary Outcome: Part A: Dose-normalized AUClast (Area Under the Concentration-Time Curve From Time 0 to Time of the Last Quantifiable Concentration) for Estimation of Relative Bioavailability for Alisertib Oral Solution (OS) Versus Powder in Capsule Formulations (PIC)
Description: Dose normalized AUClast was obtained using Cmax divided by alisertib dose in milligrams to provide values adjusted to a 1 mg alisertib dose.
Time Frame: Cycles 1 and 2 Day 1 predose and at multiple time points (up to 48 hours) postdose, and, if clinically feasible, at the time of a serious or unusual AE that was judged by the investigator to be treatment related.
Population: PK evaluable population including all participants with sufficient dosing and PK data to reliably estimate PK parameters, with data available for analysis. Data for Cycle 1 and Cycle 2 were combined for analyses.
Measure: Mean (Standard Deviation); unit: nM*hr/mg
Arm/Group | Part A: Alisertib OS | Part A: Alisertib PIC
Number analyzed (Participants) | 17 | 17
nM*hr/mg | 530.18 (177.750) | 372.53 (145.190)
Statistical Analysis 1: Comparison: Part A: Alisertib OS vs Part A: Alisertib PIC; Test type: Superiority or Other; Geometric mean ratio = 1.38, 90% CI 2-sided [1.08 to 1.78] — The CIs are calculated for the difference in the LS means of the ln-transformed Day 1 AUClast values (difference=OS-PIC). Antilogs of the confidence limits for the difference are taken to construct the CIs for the ratio of the geometric means

3. Primary Outcome: Part B: Cmax: Maximum Observed Concentration for Alisertib Administered as an Oral Solution With Food Versus Without Food
Description: Not performed.
Time Frame: as for outcome 2
Population: Data from Part B were not analyzed as planned because this part of the study was terminated after only 6 of the planned 14 PK-evaluable participants were enrolled, as the OS was not stable and gelled prior to dosing. With PK evaluability being compromised by gelling of the OS, the data were not analyzed as planned.
Groups:
- Part B: Alisertib OS (Fed State): Alisertib 35 mg (35 mg = relative bioavailability estimate in Part A as dose of OS that was calculated to yield the area under the concentration time curve of a 50-mg PIC dose): Alisertib 35 mg oral solution (OS), in fed state, once on Day 1, followed by alisertib 30 mg, OS, BID on Days 3-9, followed by a 14-day rest period in Cycle 1, in a 23-day cycle.
- Part B: Alisertib OS (Fasted State): Alisertib 35 mg, OS, in fasted state, once on Day 1, followed by alisertib 30 mg, OS, BID on Days 3-9, followed by a 14-day rest period in a 23-day cycle.
Arm/Group | Part B: Alisertib OS (Fed State) | Part B: Alisertib OS (Fasted State)
Number analyzed (Participants) | 0 | 0

4. Primary Outcome: Part B: AUClast: Area Under the Concentration-Time Curve From Time 0 to Time of the Last Quantifiable Concentration for Alisertib Administered as an Oral Solution With Food Versus Without Food
Description: Not performed.
Time Frame: as for outcome 2
Population: as for outcome 3
Arm/Group | Part B: Alisertib OS (Fed State) | Part B: Alisertib OS (Fasted State)
Number analyzed (Participants) | 0 | 0

5. Primary Outcome: Part B: Cmax: Maximum Plasma Concentration for Alisertib Oral Solution Following Multiple-Dose Administration
Description: Not performed.
Time Frame: Cycle 1 Day 9 predose and at multiple time points (up to 12 hours) postdose, and, if clinically feasible, at the time of a serious or unusual AE that was judged by the investigator to be treatment related.
Population: as for outcome 3
Arm/Group | Part B: OS Food Effect Fed/Fasted (Sequence A) | Part B: OS Food Effect Fasted/Fed (Sequence B)
Number analyzed (Participants) | 0 | 0

6. Primary Outcome: Part B: Tmax: Time of First Occurrence of Cmax Over the Dosing Interval for Alisertib Oral Solution Following Multiple-Dose Administration
Description: Not performed.
Time Frame: as for outcome 5
Population: as for outcome 3
Arm/Group | Part B: OS Food Effect Fed/Fasted (Sequence A) | Part B: OS Food Effect Fasted/Fed (Sequence B)
Number analyzed (Participants) | 0 | 0

7. Primary Outcome: Part B: AUCτ: Area Under the Concentration-Time Curve From Time 0 to End of Dosing Interval for Alisertib Oral Solution Following Multiple-Dose Administration
Description: Not performed.
Time Frame: as for outcome 5
Population: as for outcome 3
Arm/Group | Part B: OS Food Effect Fed/Fasted (Sequence A) | Part B: OS Food Effect Fasted/Fed (Sequence B)
Number analyzed (Participants) | 0 | 0

8. Primary Outcome: Part C: Cmax: Maximum Observed Concentration for Alisertib Administered as an Enteric-Coated Capsule (ECT) With Food Versus Without Food
Description: Participants were randomized to receive 50-mg alisertib as an ECT (single, 50-mg strength tablets) under fasted or fed (following a standardized high-fat meal) conditions.
Time Frame: as for outcome 2
Population: PK-evaluable population including all participants with sufficient dosing and PK data to reliably estimate PK parameters, with data available for analysis.
Measure: Mean (Standard Deviation); unit: nM
Groups:
- Part C: Alisertib ECT (Fasted State): Alisertib 50 mg, ECT, orally, in fasted state, once on Day 1, followed by alisertib 40 mg, ECT, BID on Days 3 through 9, followed by a 14-day rest period in Cycle 1 in a 23-day cycle.
- Part C: Alisertib ECT (Fed State): Alisertib 50 mg, ECT, orally, in fed state, once on Day 1, followed by alisertib 40 mg, ECT, BID on Days 3 through 9, followed by a 14-day rest period in Cycle 1 or Cycle 2.
Arm/Group | Part C: Alisertib ECT (Fasted State) | Part C: Alisertib ECT (Fed State)
Number analyzed (Participants) | 14 | 14
nM | 1757.9 (924.5) | 1401.2 (501.0)
Statistical Analysis 1: Comparison: Part C: Alisertib ECT (Fasted State) vs Part C: Alisertib ECT (Fed State); Test type: Superiority or Other; Geometric mean ratio = 0.84, 90% CI 2-sided [0.66 to 1.06] — The CIs are calculated for the difference in the LS means of the ln-transformed Day 1 Cmax values (difference=Fed-Fasted). Antilogs of the confidence limits for the difference are taken to construct the CIs for the ratio of the geometric means

9. Primary Outcome: Part C: AUClast: Area Under the Concentration-Time Curve From Time 0 to Time of the Last Quantifiable Concentration for Alisertib Administered as an Enteric-Coated Capsule (ECT) With Food Versus Without Food
Time Frame: Cycles 1 and 2 on Day 1 predose and at multiple time points (up to 48 hours) postdose, and, if clinically feasible, at the time of a serious or unusual AE that was judged by the investigator to be treatment related.
Population: The PK evaluable population including all participants with sufficient dosing and PK data to reliably estimate PK parameters, with data available for analysis.
Measure: Mean (Standard Deviation); unit: nM*h
Arm/Group | Part C: Alisertib ECT (Fasted State) | Part C: Alisertib ECT (Fed State)
Number analyzed (Participants) | 14 | 14
nM*h | 23928.6 (14343.56) | 24135.0 (11757.15)
Statistical Analysis 1: Comparison: Part C: Alisertib ECT (Fasted State) vs Part C: Alisertib ECT (Fed State); Test type: Superiority or Other; Geometric mean ratio = 1.04, 90% CI 2-sided [0.80 to 1.34] — The CIs are calculated for the difference in the LS means of the ln-transformed Day 1 AUClast values (difference=Fed-Fasted). Antilogs of the confidence limits for the difference are taken to construct the CIs for the ratio of the geometric means

10. Primary Outcome: Part C: AUC∞: Area Under the Concentration-Time Curve From Time 0 to Infinity, Calculated Using the Observed Value of the Last Quantifiable Concentration for Alisertib Administered as an Enteric-Coated Capsule (ECT) With Food Versus Without Food
Time Frame: as for outcome 9
Population: as for outcome 9
Measure: Mean (Standard Error); unit: nM*h
Arm/Group | Part C: Alisertib ECT (Fasted State) | Part C: Alisertib ECT (Fed State)
Number analyzed (Participants) | 11 | 14
nM*h | 30627.3 (21000.29) | 28507.1 (15637.50)
Statistical Analysis 1: Comparison: Part C: Alisertib ECT (Fasted State) vs Part C: Alisertib ECT (Fed State); Test type: Superiority or Other; Geometric mean ratio = 0.94, 90% CI 2-sided [0.68 to 1.32] — The CIs are calculated for the difference in the LS means of the ln-transformed Day 1 AUC values (difference=Fed-Fasted). Antilogs of the confidence limits for the difference are taken to construct the CIs for the ratio of the geometric means

11. Primary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An Adverse Event (AE) is defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment. A Serious Adverse Event (SAE) A serious is any experience that suggests a significant hazard, contraindication, side effect or precaution that: results in death, is life-threatening, required in-patient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect or is medically significant.
Time Frame: Up to 30 days after the last dose of study drug (up to 27.4 months)
Population: Safety population was defined as all participants who receive any amount of alisertib.
Measure: Number; unit: participants
Groups:
- Part A: Relative Bioavailability: Alisertib 25 or 50 mg, OS, once on Day 1, in alternating dosage in Cycles 1 and 2, followed by alisertib 40 mg PIC, orally, BID on Days 3 through 9, followed by a 14-day rest period in Cycles 1 and 2, in 23-day cycles, followed by alisertib 40-50 mg (individual dosage based on tolerability in Cycles 1 and 2), PIC, orally, BID on Days 1 through 7, followed by a 14-day rest period in Cycle 3, in 21-day cycles until disease progression, occurrence of an unacceptable alisertib-related toxicity, or the start of another anticancer therapy.
- Part B: OS Food Effect: Alisertib 35 mg (35 mg = relative bioavailability estimate in Part A as dose of OS that was calculated to yield the area under the concentration time curve of a 50-mg PIC dose), OS, once on Day 1, in alternating fed/fasted states in Cycles 1 and 2, followed by alisertib 30 mg, OS, BID on Days 3-9, followed by a 14-day rest period in Cycle 1 and 2, in 23-day cycles, followed by alisertib 40-50 mg (individual dosage based on tolerability in Cycles 1 and 2), PIC, orally, BID on Days 1-7, followed by a 14-day rest period in Cycle 3, in 21-day cycles until disease progression, occurrence of an unacceptable alisertib-related toxicity, or the start of another anticancer therapy.
- Part C: ECT Food Effect: Alisertib 50 mg, enteric-coated tablets (ECT), orally, in fed state, once on Day 1, in alternating fed/fasted states in Cycles 1 and 2, followed by alisertib 40 mg, ECT, orally, BID on Days 3 through 9, followed by a 14-day rest period in Cycle 1 and Cycle 2 in 23-day cycles, followed by alisertib 40-50 mg (individual dosage based on tolerability in Cycles 1 and 2), PIC, orally, BID on Days 1-7, followed by a 14-day rest period in Cycle 3, in 21-day cycles until disease progression, occurrence of an unacceptable alisertib-related toxicity, or the start of another anticancer therapy.
Arm/Group | Dose Escalation Cohort | Part A: Relative Bioavailability | Part B: OS Food Effect | Part C: ECT Food Effect
Number analyzed (Participants) | 4 | 19 | 6 | 24
participants
  AE | 4 | 19 | 6 | 24
  SAE | 2 | 4 | 2 | 11

12. Primary Outcome: Number of Participants With Abnormal Laboratory Values Reported as Adverse Events at an Incidence of at Least 5%
Description: Laboratory AEs reported at an incidence of at least 5% overall in the following system organ classes (SOCs) are reported: blood and lymphatic system disorders, metabolism and nutrition disorders, investigations, and hepatobiliary disorders. Abnormal laboratory value were assessed as an AE if the value leads to discontinuation or delay in treatment, dose modification, therapeutic intervention, or is considered by the investigator to be a clinically significant change from baseline. A treatment--emergent adverse event (TEAE) is defined as an adverse event with an onset that occurs after receiving study drug.
Time Frame: Up to 30 days after the last dose of study drug (up to 27.4 months)
Population: Safety Population is defined as all participants who receive any amount of alisertib.
Measure: Number; unit: participants
Arm/Group | Dose Escalation Cohort | Part A: Relative Bioavailability | Part B: OS Food Effect | Part C: ECT Food Effect
Number analyzed (Participants) | 4 | 19 | 6 | 24
participants
  Neutropenia | 3 | 8 | 2 | 21
  Leukopenia | 3 | 7 | 2 | 17
  Anaemia | 3 | 4 | 2 | 15
  Thrombocytopenia | 4 | 3 | 3 | 10
  Lymphopenia | 0 | 3 | 0 | 3
  Hypomagnesaemia | 0 | 0 | 1 | 7
  Hyperglycaemia | 0 | 1 | 1 | 3
  Hypokalaemia | 0 | 0 | 1 | 3
  White blood cell count decreased | 0 | 0 | 1 | 5
  Aspartate aminotransferase increased | 1 | 0 | 0 | 6
  Gamma-glutamyltransferase increased | 0 | 1 | 0 | 2
  Lymphocyte count decreased | 0 | 0 | 0 | 3
  Neutrophil count decreased | 0 | 1 | 0 | 2
  Hyperbilirubinaemia | 1 | 0 | 0 | 3

13. Primary Outcome: Number of Participants With Abnormal Vital Signs Reported as Adverse Events
Description: Vital signs (blood pressure, heart rate, and oral temperature) measurements were obtained throughout the study.
Time Frame: Up to 30 days after the last dose of study drug (up to 24 months approximately)
Population: Safety Population is defined as all participants who receive any amount of alisertib.
Measure: Number; unit: participants
Arm/Group | Dose Escalation Cohort | Part A: Relative Bioavailability | Part B: OS Food Effect | Part C: ECT Food Effect
Number analyzed (Participants) | 4 | 19 | 6 | 24
participants
  Hypertension | 1 | 0 | 1 | 1
  Hypotension | 0 | 1 | 1 | 0
  Tachycardia | 1 | 1 | 1 | 0
  Sinus bradycardia | 0 | 0 | 0 | 1

14. Secondary Outcome: Best Overall Response (CR+PR) Based on Investigator's Assessment According to the Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1
Description: Best overall response is defined as the number of participants with Complete Response (CR) + Partial Response (PR) as assessed by the investigator according to Response Evaluation Criteria in Solid Tumors (RECIST) criteria 1.1 for target lesions and assessed by CT or MRI. CR is defined as disappearance of all target lesions and PR is defined as 30% decrease in the sum of the longest diameter (LD) of target lesions. Stable Disease (SD) is defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for Progressive Disease, taking as reference the smallest sum LD since the treatment started.
Time Frame: At the completion of Cycle 2 and every 2 cycles (every 6 weeks) until Cycle 6 (18 weeks). After Cycle 6 (18 weeks), CT/MRI scans (with contrast) were to be performed every 3 cycles (9 weeks) until PD was documented.
Population: Efficacy analysis included all participants who had a baseline response assessment and at least one on-study response assessment.
Measure: Number; unit: participants
Arm/Group | Dose Escalation Cohort | Part A: Relative Bioavailability OS/PIC (Sequence A) | Part A: Relative Bioavailability PIC/OS (Sequence B) | Part B: OS Food Effect Fed/Fasted (Sequence A) | Part B: OS Food Effect Fasted/Fed (Sequence B) | Part C: ECT Food Effect Fed/Fasted (Sequence A) | Part C: ECT Food Effect Fasted/Fed (Sequence B)
Number analyzed (Participants) | 2 | 8 | 9 | 3 | 3 | 12 | 12
participants
  Best Overall Response of CR or PR | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Best Overall Response of Stable Disease | 0 | 1 | 5 | 2 | 1 | 6 | 6

ADVERSE EVENTS:
Time Frame: Up to 30 days after the last dose of study drug (up to 27.4 months approximately)
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Dose Escalation Cohort | Part A: Relative Bioavailability | Part B: OS Food Effect | Part C: ECT Food Effect
Serious Adverse Events (participants affected / at risk) | 2/4 | 4/19 | 2/6 | 11/24
Other Adverse Events (participants affected / at risk) | 4/4 | 19/19 | 6/6 | 24/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dose Escalation Cohort (N=4) | Part A: Relative Bioavailability (N=19) | Part B: OS Food Effect (N=6) | Part C: ECT Food Effect (N=24)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 1 | 2
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Fatigue (General disorders) | 0 | 0 | 1 | 0
Pain (General disorders) | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Anuria (Renal and urinary disorders) | 0 | 0 | 0 | 1
Hydronephrosis (Renal and urinary disorders) | 0 | 1 | 0 | 1
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 — One treatment-emergent death occurred during treatment with alisertib and is not related.
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Female genital tract fistula (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 0 | 1
Bile duct stone (Hepatobiliary disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dose Escalation Cohort (N=4) | Part A: Relative Bioavailability (N=19) | Part B: OS Food Effect (N=6) | Part C: ECT Food Effect (N=24)
Diarrhoea (Gastrointestinal disorders) | 0 | 11 | 1 | 13
Nausea (Gastrointestinal disorders) | 2 | 10 | 2 | 9
Stomatitis (Gastrointestinal disorders) | 4 | 7 | 5 | 6
Vomiting (Gastrointestinal disorders) | 0 | 7 | 1 | 5
Constipation (Gastrointestinal disorders) | 0 | 1 | 1 | 6
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 1 | 3
Abdominal distension (Gastrointestinal disorders) | 1 | 1 | 0 | 3
Dysphagia (Gastrointestinal disorders) | 0 | 2 | 1 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0 | 2
Flatulence (Gastrointestinal disorders) | 0 | 1 | 1 | 1
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Ascites (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Ileus (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 2 | 8 | 2 | 17
Leukopenia (Blood and lymphatic system disorders) | 3 | 7 | 2 | 13
Anaemia (Blood and lymphatic system disorders) | 3 | 4 | 2 | 13
Thrombocytopenia (Blood and lymphatic system disorders) | 4 | 3 | 3 | 7
Lymphopenia (Blood and lymphatic system disorders) | 0 | 3 | 0 | 3
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 5 | 1 | 13
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 2 | 1 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2
Palmar erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1
Pruritus generalised (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Papule (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Rash generalised (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Skin disorder (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Fatigue (General disorders) | 3 | 12 | 4 | 11
Asthenia (General disorders) | 1 | 2 | 1 | 3
Pyrexia (General disorders) | 2 | 2 | 2 | 1
Oedema peripheral (General disorders) | 1 | 2 | 0 | 1
Early satiety (General disorders) | 0 | 0 | 1 | 1
Chest discomfort (General disorders) | 0 | 1 | 0 | 0
Mucosal inflammation (General disorders) | 0 | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 2 | 7 | 1 | 7
Dehydration (Metabolism and nutrition disorders) | 0 | 2 | 0 | 4
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 5
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 3
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1
Gout (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Oral candidiasis (Infections and infestations) | 1 | 2 | 2 | 4
Sinusitis (Infections and infestations) | 0 | 2 | 0 | 2
Upper respiratory tract infection (Infections and infestations) | 0 | 2 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 2
Nasopharyngitis (Infections and infestations) | 0 | 1 | 0 | 1
Oral herpes (Infections and infestations) | 0 | 1 | 0 | 1
Clostridium difficile infection (Infections and infestations) | 1 | 0 | 0 | 0
Fungal skin infection (Infections and infestations) | 0 | 1 | 0 | 0
Herpes simplex (Infections and infestations) | 1 | 0 | 0 | 0
Skin infection (Infections and infestations) | 0 | 1 | 0 | 0
Vaginal infection (Infections and infestations) | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 6 | 0 | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 4 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0
Axillary mass (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 2 | 2 | 0 | 4
Somnolence (Nervous system disorders) | 0 | 2 | 0 | 2
Dizziness (Nervous system disorders) | 1 | 2 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 2 | 0 | 1
Cognitive disorder (Nervous system disorders) | 2 | 0 | 0 | 0
Memory impairment (Nervous system disorders) | 0 | 2 | 0 | 0
Balance disorder (Nervous system disorders) | 1 | 0 | 0 | 0
Brain oedema (Nervous system disorders) | 0 | 1 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 1 | 0
Nerve compression (Nervous system disorders) | 0 | 1 | 0 | 0
Weight decreased (Investigations) | 0 | 3 | 0 | 5
White blood cell count decreased (Investigations) | 0 | 0 | 1 | 5
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 0 | 4
Gamma-glutamyltransferase increased (Investigations) | 0 | 1 | 0 | 2
Neutrophil count decreased (Investigations) | 0 | 1 | 0 | 2
Alanine aminotransferase increased (Investigations) | 0 | 1 | 0 | 1
Blood urea increased (Investigations) | 0 | 0 | 0 | 2
Lymphocyte count decreased (Investigations) | 0 | 0 | 0 | 2
Blood phosphorus decreased (Investigations) | 0 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Depression (Psychiatric disorders) | 0 | 2 | 0 | 2
Anxiety (Psychiatric disorders) | 0 | 1 | 1 | 1
Confusional state (Psychiatric disorders) | 0 | 1 | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 1 | 0 | 1
Delirium (Psychiatric disorders) | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 1 | 0 | 1 | 2
Hypotension (Vascular disorders) | 0 | 1 | 1 | 0
Raynaud's phenomenon (Vascular disorders) | 0 | 0 | 0 | 2
Vision blurred (Eye disorders) | 1 | 0 | 1 | 0
Diplopia (Eye disorders) | 0 | 1 | 0 | 0
Eyelid pain (Eye disorders) | 0 | 1 | 0 | 0
Lacrimation increased (Eye disorders) | 0 | 1 | 0 | 0
Visual impairment (Eye disorders) | 0 | 1 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0 | 0 | 3
Jaundice (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Tachycardia (Cardiac disorders) | 1 | 1 | 1 | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 1 | 0 | 2
Vulvovaginal pruritus (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Forearm fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Tumour flare (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 0 | 0 | 1 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 1 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In general, Investigators may publish clinical data after the earlier of (i) publication by the Sponsor or (ii) 12 months following the abandonment, early termination or database lock; provided a copy of the publication provided to Sponsor at least 30 days ahead of publication, the Sponsor's confidential information is removed as may be requested by Sponsor and Investigator defers publication for up to 60 days in the event Sponsor provides notice that it intends to file a patent application.